CLINICAL TRIAL: NCT01746056
Title: A Comparative Study of Occlusive Heat Patch Vs. No Treatment in the Treatment of Verruca
Brief Title: A Comparative Study of Occlusive Heat Patch in the Treatment of Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Ferndale Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1209010850
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Verruca (Warts)
Keywords: Warts; Verruca; Heat patch
MeSH Terms: conditions — Warts

STUDY DESIGN:
Intervention Model Description: one arm receiving intervention in daily for 12 week the other receives the intervention 2 weeks on and 2 weeks off for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Heat Patch Continuous (Active Comparator): applied 2 hrs daily for 12 weeks
  Interventions: Device: Occlusive Heat Patch
- Heat Patch Noncontinuous (Active Comparator): applied 2 hrs daily 2 weeks on and 2 weeks off for 12 weeks
  Interventions: Device: Occlusive Heat Patch

INTERVENTIONS:
Device: Occlusive Heat Patch — The heat patch will be applied for 2 hours every day for a period of 12 weeks.

SUMMARY:
The goal of this study is to determine the safety and efficacy of the occlusive heat patch for the treatment of verrucae (warts).

DETAILED DESCRIPTION:
Human papillomavirus (HPV) is a virus that causes verrucae, or warts, on the skin, particularly of the distal extremities, and lesions of the mucous membranes. Warts are highly prevalent, occurring in up to 13% of the general population and in around 25% of otherwise healthy children. About 67% of warts resolve spontaneously within two years; however more than 25% will persist for many years, some resulting in pain or dysfunction and some imparting significant psychosocial problems. Localized hyperthermia (warming) has been reported to be effective in the treatment of HPV-induced warts for nearly two decades. A novel method of treating warts with heat is the use of an occlusive patch that contains a mixture of chemicals (ferric chloride), which in the presence of oxygen reacts to generate reproducible thermal warming of the skin to a temperature of 42-43ºC for at least two hours. The heat is believed to alter the immune response and kill the HPV virus in the wart tissue.

The changes to the title, endpoints, inclusion and exclusion criteria were revised to reflect the second, final phase of this trial. The first portion of the trial, a proof of concept trial, was completed and the results published in an article added to the citations section.

A significant delay occurred in completion of this second phase of the trial due to personnel issues and interruptions secondary to COVID-19 pandemic restrictions.

ELIGIBILITY:
Inclusion Criteria:

Proof of Concept Study:

* Male or non-pregnant female 5 years of age or older.
* Written consent (adults) and written assent (minors).
* Subjects with a minimum of two clinically diagnosed verrucae 4 cm in diameter or less in a similar treatment area.
* Subjects must be willing and able to apply the occlusive heat patch(s) as directed, comply with study instructions and return to the clinic for required visits.
* Women of childbearing potential (WOCBP) must agree to use an effective form of birth control for the duration of the study (abstinence, stabilized on oral contraceptives or contraceptive patches for at least three months, implant, injection, intrauterine device, NuvaRing®, condom and spermicidal or diaphragm and spermicidal). Abstinence is an acceptable form of birth control for subjects who are not sexually active. Subjects that become sexually active during the trial must agree to use an effective, non-prohibited form of birth control for the duration of the study.

Confirmation Study:

* Male or female 5 -25 years of age at the baseline visit.
* Written consent (adults) and written assent (minors).
* Subjects with one clinically diagnosed verruca, 2-20 mm in largest diameter.
* Subjects must be willing and able to apply the study patch as directed, comply with study instructions and return for required visits.

Exclusion Criteria:

Proof of Concept Study:

* Subjects who are immunocompromised for any reason or are known to be HIV+ based on medical history taken at screening.
* Subjects taking any of the following systemic therapy with 4 weeks of enrollment; cimetidine, systemic steroids, immunomodulators or immunosuppressants.
* Subjects who have used any anti-verruca treatments within 4 weeks. These include but are not limited to topical salicylic acid preparations, imiquimod (Aldara), podophyllin containing preparations, surgical procedures, immunotherapy, among others.
* Subjects who have active localized or systemic medical conditions that in the opinion of the investigator, would preclude their participation in the study or interfere with their assessment of their verrucae.
* Subjects with any underlying disease(s) or a dermatological condition of the affected area(s) that requires the use of interfering topical or systemic therapy.
* Subjects with verruca, for treatment, that are located in the periungual, genital, or head regions or have mosaic warts.
* Subjects with verruca, for treatment, that is associated with significant scarring from prior therapy in the opinion of the investigator.
* Subjects who are unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function.
* Subjects with any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in a research study.
* Subjects with a history of allergy or sensitivity to any of the components or the patches (including the adhesives).
* Subjects who are currently enrolled in a clinical drug or device research study.
* Subjects who have been treated with another investigational device or drug within 30 days prior to study enrollment.
* Subject is pregnant, nursing or planning a pregnancy during the study period

Confirmation Study:

* Subjects who are immunocompromised for any reason or are known to be HIV+ based on medical history taken at screening.
* Subjects taking any of the following systemic therapy within 4 weeks of enrollment; cimetidine, systemic steroids, immunomodulators or immunosuppressants.
* Subjects who have used any destructive anti-verruca treatments within 4 weeks. These include but are not limited to cryotherapy, topical salicylic acid preparations, podophyllin-containing preparations, intralesional bleomycin, or surgical procedures. No immunotherapy (topical allergens or intralesional antigen injections) or topical sinecatechins ointment, imiquimod cream 6 months before baseline visit.
* Subjects who have active localized or systemic medical conditions that in the opinion of the investigator, would preclude their participation in the study or interfere with their assessment of their verrucae.
* Subjects with any underlying disease(s) or a dermatological condition of the affected area(s) that requires the use of interfering topical or systemic therapy.
* Subjects with verrucae only located in the genital or head regions or possessing only mosaic, flat or filiform warts.
* Subjects with verrucae only located in areas with significant scarring from prior therapy in the opinion of the investigator.
* Subjects who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
* Subjects with any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in a research study.
* Subjects with a history of allergy or sensitivity to any of the components of the patches (including the liquid adhesive and adhesive remover).
* Subjects who are currently enrolled in a clinical drug or device research study.
* Subjects who have been treated with another investigational device or drug within 30 days prior to study enrollment.
* Subject is pregnant, nursing or planning a pregnancy during the study period.
* During the study, concomitant use of the following medications or treatments is PROHIBITED:

  * Systemic corticosteroids, immunosuppressants, immunomodulators, cimetidine. Topical treatments to the area containing the target verruca intended to treat warts including, podophyllin, salicylic acid preparations, intralesional bleomycin, surgical procedures or immunotherapy (topical allergens or intralesional antigen injections) or topical sinecatechins ointment and imiquimod cream among others.
  * Medications or treatments that might interfere with the evaluation of the occlusive patch should not be used.
  * Changes in general skin care treatment during the study should also be discouraged.
  * There will be no use of medication which, in the opinion of the investigators, will interfere with the study results.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-12; Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Percent reduction in verrucae diameter - proof of concept study | 12 weeks
  Efficacy will be determined by the percent reduction in verruca diameter (Lesion Measurement). A severity grade will be given to the target and control warts using the Investigator Global Improvement Score (IGIS). IGIS scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score = 0 on target verruca - confirmation study | 24 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects (in each arm and combined) achieving an IGIS of 0 (complete clearance) of the target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score = 0 on at least 1 non-target verruca - confirmation study | 24 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects greater than one verruca that demonstrate clearance of one or more than one non-target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.

SECONDARY OUTCOMES:
Count of participants with an IGS score = 0 on target verruca - confirmation study | 12 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects (in each arm and combined) achieving an IGIS of 0 (complete clearance) of the target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score = 0 on target verruca - confirmation study | 36 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects (in each arm and combined) achieving an IGIS of 0 (complete clearance) of the target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score = 0 on at least 1 non-target verruca - confirmation study | 12 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects greater than one verruca that demonstrate clearance of one or more than one non-target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score = 0 on at least 1 non-target verruca - confirmation study | 36 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects greater than one verruca that demonstrate clearance of one or more than one non-target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score < = 2 on target verruca - confirmation study | 12 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects (in each arm and combined) achieving an IGIS of < = 2 of the target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score < = 2 on target verruca - confirmation study | 24 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects (in each arm and combined) achieving an IGIS of < = 2 of the target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score < = 2 on target verruca - confirmation study | 36 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects (in each arm and combined) achieving an IGIS of < = 2 of the target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score < = 2 on at least 1 non-target verruca - confirmation study | 12 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects greater than one verruca that demonstrate an IGS score < = 2 on one or more non-target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score < = 2 on at least 1 non-target verruca - confirmation study | 24 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects greater than one verruca that demonstrate an IGS score < = 2 on one or more non-target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.
Count of participants with an IGS score < = 2 on at least 1 non-target verruca - confirmation study | 36 weeks
  To assess the efficacy of the heat patch in the confirmation study, the count of subjects greater than one verruca that demonstrate an IGS score < = 2 on one or more non-target verruca will be assessed. Investigator Global Improvement Score (IGIS) scale scores are as follows: 4 = Same or worse, 3 = Minimal Improvement, 2 = Marked Improvement, 1 = Almost Clear, 0 = Clear.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Antaya, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Result] Antaya RJ, del Carmen M, Alonso F, Sukumar N, Yong F, Dvoretzky I. An Open Label Study of an Occlusive Heat Patch in the Treatment of Warts. J Drugs Dermatol. 2019 Apr 1;18(4):368-373. PMID 31012566